CLINICAL TRIAL: NCT01853670
Title: Kilovoltage Conebeam Imaging Based Adaptive Radiation Therapy for Head & Neck Patients Treated With Intensity Modulated Radiation Therapy
Brief Title: Adaptive Radiation Therapy for Head & Neck Cancer Patients
Acronym: IGRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167-08
Record Dates: First submitted 2013-02-25; First posted 2013-05-15 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-09

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- definitive radiation + concomitant chemo (Experimental): Concurrent chemo + IGRT:
  These patients will have chemotherapy during the time of radiation treatment
  Interventions: Radiation: concurrent chemo + IGRT
- neoadjuvant chemo (Experimental): Neoadjuvant chemo + IGRT:
  These patients will have chemotherapy prior to other radiation treatment.
  Interventions: Radiation: neoadjuvant chemo + IGRT

INTERVENTIONS:
Radiation: concurrent chemo + IGRT
  Arms: definitive radiation + concomitant chemo
Radiation: neoadjuvant chemo + IGRT
  Arms: neoadjuvant chemo

SUMMARY:
The purpose of this study is to determine the utility of kilovoltage (kV) cone beam CT imaging to track the dose delivered in head and neck cancer patients, to assess the benefit of cone beam CT to patients set-up for radiation treatment, to determine how shifts based on kV cone beam CT compare to the standard approach (orthogonal pair), and to develop remote access tools (preferably internet-based) so that the MD can approve these plans in real time.

DETAILED DESCRIPTION:
The investigators' secondary objectives for this study are to assess the possibility of using kV cone beam for treatment replanning as compared to standard the treatment planning, to determine the need and feasibility of adaptive radiation therapy, to develop concept of establishing cumulative DVH (C-DVH) with daily updates and compare it to planned DVH (P-DVH), to identify tolerance margins, to evaluate local control, locoregional control, distant metastasis, and overall survival, to assess patient quality of life,and to develop predictors of patients which may benefit from ART.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have an ECOG (Eastern Clinical Oncology Group) performance status of 0-2
* Patients should meet at least one of the following criteria:

  1. Locally advanced cancer (T3-T4 and/or N2-N3)
  2. Tumors wrapping around critical structures such as the optic nerves, optic chiasm, or brainstem
  3. Significant expected weight loss.

Exclusion Criteria:

* Previous surgical procedure more significant than a biopsy to the primary tumor or regional lymph nodes.
* Poor renal function (inability to undergo a CT with IV contrast)
* Previous radiation therapy to the head and neck.
* Inability to tolerate prolonged immobilization.
* Children and women who are pregnant or decline to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical patient response | From the date of initiation of radiation therapy, until date of first progression or until date of death (approximately 5 years).
  This will assessed by CT scan or MRI 4-5 weeks post concurrent chemo.

SECONDARY OUTCOMES:
Patient quality of life | During radiation therapy (7-9 weeks)
  This will be assessed using the: Fact Head & Neck form at baseline, and weekly throughout radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Hu, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States